CLINICAL TRIAL: NCT00695630
Title: Flumazenil Rescue Strategy
Brief Title: Flumazenil Reversal of Oral Triazolam
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Peter Milgrom/Professor of Dental Public Health Sciences, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 30779; U54DE014254 (NIH); T32007132
Record Dates: First submitted 2008-06-09; First posted 2008-06-12 (Estimated); Last update posted 2008-06-12 (Estimated); Status verified 2008-06

CONDITIONS: Dental Anxiety
Keywords: conscious sedation; dental anxiety/drug therapy; behavior/drug effects
MeSH Terms: interventions — Flumazenil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Flumazenil 2mL
  Interventions: Drug: Flumazenil
- 2 (Placebo Comparator): Saline, 2mL SM
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Flumazenil — 2 mL, 0.2 mg SM
  Arms: 1
Drug: Placebo — 2 mL sterile saline SM
  Arms: 2

SUMMARY:
An increase in the utilization of anesthesia and sedation medications by non-anesthesiologists, including dentists, has grown dramatically. This has been prompted, in part, by the need for pharmacological tools to address high levels of fear and anxiety about dental care among the US population and the evidence of oral health disparities among those who are fearful . Given the prevalence of dental fear in the general population and in the various populations with the greatest burden of oral diseases, effective sedation techniques are needed that are safe and effective in the hands of general dentists that make up the "front line" in the efforts to reduce oral health disparities. This study is to determine whether, when compared to a saline placebo, a single intraoral submucosal administration of the benzodiazepine antagonist flumazenil (0.2 mg) is capable of attenuating in 10 minutes or less the central nervous system (CNS) depression produced by a paradigm of stacked sublingual dosing of triazolam (3 doses of 0.25 mg over 90 minutes).

ELIGIBILITY:
Inclusion Criteria:

* ASA I

Exclusion Criteria:

* Use of benzodiazepines, anxiolytics or any other medications that would interact with either triazolam's or flumazenil's metabolism or clinical effect (including herbals) within four weeks of the study
* Body mass index (BMI) no less than 15 kg/m2 and no greater than 30 kg/m2
* Pregnancy or not currently using pharmacologic methods of birth control
* Allergy or sensitivity to benzodiazepines
* History of a seizure disorder; AND
* Chronic tobacco use.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2006-09; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Observer Assessment of Alertness/Sedation | 360 minutes

SECONDARY OUTCOMES:
BIS | 360 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Peter M Milgrom, DDS, Principal Investigator — University of Washington
Locations (1):
- Dental Fears Research Clinic, Seattle, Washington, United States

REFERENCES:
- [Background] Jackson DL, Milgrom P, Heacox GA, Kharasch ED. Pharmacokinetics and clinical effects of multidose sublingual triazolam in healthy volunteers. J Clin Psychopharmacol. 2006 Feb;26(1):4-8. doi: 10.1097/01.jcp.0000186742.07148.da. PMID 16415697